CLINICAL TRIAL: NCT04934228
Title: Mitigating the Pro-inflammatory Phenotype of Obesity
Acronym: MAPLE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Seth Holwerda PhD, Principal Investigator, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 00147099
Record Dates: First submitted 2021-03-31; First posted 2021-06-22 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Blood Pressure; Diabetes; Obesity; Insulin Resistance; Diuretics Drug Reactions; Sympathetic Nerve Activity
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Insulin Resistance | interventions — Hydrochlorothiazide; Clonidine

STUDY DESIGN:
Intervention Model Description: Mixed Model ANOVA 3-way analysis of variance to assess pain and BP responses to the clonidine, diuretic vs. placebo.
Who Masked: Participant, Investigator
Masking Description: Randomized, double-blinded, parallel-design approach. Randomization to either the clonidine, diuretic vs. placebo will occur determined/generated by computer generated randomization and stratified by age and sex to balance the three groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): KU Investigational Pharmacy will provide the drug prescription bottle with 35-day supply of placebo to the research coordinator to give to the research participant.
  The placebo is an inert substance with no intended medical value and is used as a negative control for comparison with the study drug.
  Participants will receive a Placebo Pill; has no active ingredients but is made to look like the study drug.
  Interventions: Drug: Placebo
- Clonidine (Experimental): KU Investigational Pharmacy will provide the drug prescription bottle with 35-day supply of clonidine to the research coordinator to give to the research participant.
  Planned use in this study
  1. Condition/disease indication(s): Vascular function and blood flow
  2. Subject population: Hypertension
  3. Dose(s): 0.1 mg (oral)
  4. Administration: Oral
  5. Dosing regimen: 0.1 mg twice daily by mouth
  Interventions: Drug: Clonidine Pill
- Hydrochlorothiazide (HCTZ) (Experimental): KU Investigational Pharmacy will provide the drug prescription bottle with 35-day supply of Hydrochlorothiazide to the research coordinator to give to the research participant.
  Planned use in this study
  1. Condition/disease indication(s): Hypertension
  2. Subject population: Hypertension
  3. Dose(s): 25 mg/day
  4. Administration: Oral
  5. Dosing regimen: 12.5 mg twice per day
  Interventions: Drug: Hydrochlorothiazide 12.5Mg Tab

INTERVENTIONS:
Drug: Hydrochlorothiazide 12.5Mg Tab — Will receive 4 week supply (35 days) of Hydrochlorothiazide Pills (12.5 mg twice a day)
  Planned use in this study
  1. Condition/disease indication(s): Hypertension
  2. Subject population: Hypertension
  3. Dose(s): 25 mg/day
  4. Administration: Oral
  5. Dosing regimen: 12.5 mg twice per day
  Other Names: Hydrochlorothiazide
  Arms: Hydrochlorothiazide (HCTZ)
Drug: Clonidine Pill — Will receive 4 week supply (35 days) of Clonidine Pills (0.1 mg twice/day)
  Planned use in this study
  1. Condition/disease indication(s): Vascular function and blood flow
  2. Subject population: Hypertension
  3. Dose(s): 0.1 mg (oral)
  4. Administration: Oral
  5. Dosing regimen: 0.1 mg twice daily by mouth
  Other Names: Clonidine
  Arms: Clonidine
Drug: Placebo — Will receive a 4 week supply (35 days) of Placebo Pills; has no active ingredients but is made to look like the study drug.
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the hypothesize that 4 weeks of sympathetic nerve activity (SNA) inhibition (oral clonidine) will cause a significant reduction in circulating blood concentrations and endothelial cell expression of inflammatory markers (e.g., TNF-α, IL-6).

Our study is a prospective study using a randomized, double-blinded design to test 4 weeks of SNA blockade (oral clonidine) compared with a BP-lowering control condition (diuretic, hydrochlorothiazide) or a placebo.

DETAILED DESCRIPTION:
1. Using a randomized, double-blinded, parallel-design approach, we hypothesize that 4 weeks of SNA blockade (oral clonidine) will cause a significant reduction in expression of inflammatory markers in blood, endothelial cells, and central adipose compared with a BP-lowering control condition using hydrochlorothiazide (HCTZ) and a separate placebo treatment.
2. Determine the extent to which inflammation in the body is caused by elevated sympathetic nerve activity

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, age 18-79
* Obese: BMI > 30 m/kg2
* Hypertensive: blood pressure >130/80
* Elevated insulin resistance (HOMA-IR > 2.5)
* Waist circ: >102 cm (men) and >88 cm (women)
* Fasting glucose < 126 mg/dL
* Fasting triglycerides < 250 mg/dL
* HbA1c < 6.5%
* Willing to visit research lab (Fairway CTSU)
* Willing to undergo a blood draw
* Able to provide written informed consent

Exclusion Criteria:

* Current use of clonidine or beta-blockers
* Current smoker or History of smoking in the past 3 months.
* Hyperlipidemia: Fasting triglycerides > 250 mg/dL
* Currently taking hypertension medication
* History of heart disease (e.g., myocardial infarction, stent, byass, heart attack, stroke, heart failure, valvular heart disease, cardiomyopathy)
* History of neurological disorders
* History of transplant
* Actively participating in other studies, except for a registry study.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Blood Work: Efficacy of 4-week supply of Clonidine Compared VS 4-week supply of control condition using hydrochlorothiazide (HCTZ) and a separate placebo treatment | Baseline
  Difference in inflammatory markers in blood compared with a BP-lowering control condition using hydrochlorothiazide (HCTZ) and a separate placebo treatment
  * Norepinephrine (inflammation) Blood Test: pg/mL normal range for norepinephrine is 70 to 1700 pg/mL
  * Tumor necrosis factor-alpha (TNF-α) and interlukin-6 (IL6) Blood Test: pg/mL normal values: IL-6 was 6-31 pg/mL and TNF-α 5 pg/mL,
  * Nitrotyrosine (Oxidative stress)
Endothelial Cell Sample: Efficacy of 4-week supply of Clonidine Compared VS 4-week supply of control condition using hydrochlorothiazide (HCTZ) and a separate placebo treatment | Baseline
  Difference in endothelial cells samples compared with a BP-lowering control condition using hydrochlorothiazide (HCTZ) and a separate placebo treatment
  Endothelial cell tissue will be assessed by the KU Histology Core for markers of inflammation and oxidative stress independently from the PI's lab,
Adipose Tissue Sample: Efficacy of 4-week supply of Clonidine Compared VS 4-week supply of control condition using hydrochlorothiazide (HCTZ) and a separate placebo treatment | Baseline
  Difference in central adipose compared with a BP-lowering control condition using hydrochlorothiazide (HCTZ) and a separate placebo treatment
  Adipose tissue are expected following 4 weeks of clonidine but not HCTZ or placebo
Blood Work: Efficacy of 4-week supply of Clonidine Compared VS 4-week supply of control condition using hydrochlorothiazide (HCTZ) and a separate placebo treatment | 1 Week
  The difference in electrolytes blood test of participants in the Clonidine group compared with a BP-lowering control condition using hydrochlorothiazide (HCTZ) and a separate placebo treatment.
  • Blood Test: Electrolyte check by examining potassium concentration in blood. If potassium is 3.5 millimoles per liter or lower, oral 10 mg KCL will be prescribed to subject by a physician.
Blood Work: Efficacy of 4-week supply of Clonidine Compared VS 4-week supply of control condition using hydrochlorothiazide (HCTZ) and a separate placebo treatment | 2 Week
  The difference in electrolytes blood test of participants in the Clonidine group compared with a BP-lowering control condition using hydrochlorothiazide (HCTZ) and a separate placebo treatment.
  • Blood Test: Electrolyte check by examining potassium concentration in blood. If potassium is 3.5 millimoles per liter or lower, oral 10 mg KCL will be prescribed to subject by a physician.
Blood Work: Efficacy of 4-week supply of Clonidine Compared VS 4-week supply of control condition using hydrochlorothiazide (HCTZ) and a separate placebo treatment | 4 Week
  Difference in inflammatory markers in blood, endothelial cells, and central adipose compared with a BP-lowering control condition using hydrochlorothiazide (HCTZ) and a separate placebo treatment
  * Norepinephrine (inflammation) Blood Test: pg/mL normal range for norepinephrine is 70 to 1700 pg/mL
  * Tumor necrosis factor-alpha (TNF-α) and interlukin-6 (IL6) Blood Test: pg/mL normal values: IL-6 was 6-31 pg/mL and TNF-α 5 pg/mL,
  * Nitrotyrosine (Oxidative stress)
Endothelial Cell Sample: Efficacy of 4-week supply of Clonidine Compared VS 4-week supply of control condition using hydrochlorothiazide (HCTZ) and a separate placebo treatment | 4 Week
  Difference in endothelial cells samples compared with a BP-lowering control condition using hydrochlorothiazide (HCTZ) and a separate placebo treatment
  Endothelial cell tissue will be assessed by the KU Histology Core for markers of inflammation and oxidative stress independently from the PI's lab,
Adipose Tissue Sample: Efficacy of 4-week supply of Clonidine Compared VS 4-week supply of control condition using hydrochlorothiazide (HCTZ) and a separate placebo treatment | 4 Week
  Difference in central adipose compared with a BP-lowering control condition using hydrochlorothiazide (HCTZ) and a separate placebo treatment
  Adipose tissue are expected following 4 weeks of clonidine but not HCTZ or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Seth W. W Holwerda, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No